CLINICAL TRIAL: NCT00582205
Title: Feasibility Trial of Intraperitoneal Chemotherapy in Stage IA, IB, IC, II, III, IV and Recurrent Platinum Sensitive Ovarian, Fallopian Tube, and Primary Peritoneal Carcinoma and Stage III and IV Uterine Cancer
Brief Title: Feasibility Trial of Intraperitoneal Chemotherapy for Ovarian, Fallopian Tube, and Primary Peritoneal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study completed per investigator.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WalkerIP
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Uterine Cancer
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Uterine Cancer; Intraperitoneal Chemotherapy; IP Chemotherapy; Gynecologic Cancer; Women's Cancer; Cisplatin; Paclitaxel; Recurrent Platinum Sensitive Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Uterine Neoplasms | interventions — TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel, Cisplatin IP (Experimental): There is only one arm for this study and it represents the participants receiving the intraperitoneal chemotherapy
  Interventions: Drug: Paclitaxel, Cisplatin IP

INTERVENTIONS:
Drug: Paclitaxel, Cisplatin IP — Paclitaxel 135 mg/m2 IV (3-hr infusion) on Day 1, Cisplatin 50 mg/m2 IP on Days 1 and 8, Repeat every 3 weeks for 6 cycles

SUMMARY:
The purpose of this study is to evaluate giving chemotherapy drugs directly into the abdomen (belly) along with intravenous administration.

DETAILED DESCRIPTION:
Giving chemotherapy directly into the abdomen is called intraperitoneal (IP) chemotherapy. Because ovarian, fallopian, primary peritoneal and uterine cancer spread in the abdominal cavity, giving chemotherapy drugs by infusion into the abdominal cavity may result in a greater dose of the drugs reaching the tumor cells. Intraperitoneal treatments will be administered through an implantable peritoneal catheter. These catheters are to be inserted into the peritoneal cavity, tunneled through the subcutaneous tissue, and connected to an implantable port, which is placed in the subcutaneous tissue of the anterior, inferior thorax.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IA, IB, IC, II, III, IV and recurrent platinum sensitive epithelial ovarian carcinoma, fallopian tube carcinoma, primary peritoneal carcinoma, or ovarian carcinosarcoma. Histologic subtypes which are eligible include serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's tumor, adenocarcinoma (not otherwise specified), and carcinosarcoma.
* Patients with advanced endometrial carcinoma, of any histology, including endometrioid adenocarcinoma, clear cell adenocarcinoma, and serous papillary carcinoma.
* Patients with uterine carcinosarcoma of any stage are eligible.

Exclusion Criteria:

* Patients with epithelial ovarian carcinoma of low malignant potential (borderline carcinomas).
* Patients with septicemia, severe infection, or acute hepatitis.
* Patients with prior malignancy or cancer treatment within the last five years.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Walker, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paclitaxel, Cisplatin IP
Started | 21
Completed | 11
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel, Cisplatin IP
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 61 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Are Able to Receive 6 Cycles of Intraperitoneal Cisplatin Chemotherapy.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel, Cisplatin IP
Number analyzed (Participants) | 21
Participants | 7

2. Secondary Outcome: Number of Patients With Dose Reductions or Dose Delays Due to Neuropathy or Toxicity
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel, Cisplatin IP
Number analyzed (Participants) | 17
Participants | 7

ADVERSE EVENTS:
Arm/Group | Paclitaxel, Cisplatin IP
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel, Cisplatin IP (N=21)
small bowel obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel, Cisplatin IP (N=21)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) — Resulting in dose delays

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes